CLINICAL TRIAL: NCT02647970
Title: Stearoyl-CoA Desaturase and Energy Metabolism in Humans
Acronym: SEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: The Research Council of Norway (Other); University of Oxford (Other)
Responsible Party: Principal Investigator, Kathrine Vinknes, PhD, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 239948-A; 2015/634 (Other: South-Eastern Norway Regional Health Authority)
Record Dates: First submitted 2015-12-04; First posted 2016-01-06 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Healthy; Obesity
Keywords: Energy metabolism
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Dietary intervention
  Interventions: Behavioral: PUFA-Cys/Met diet
- Group B (Active Comparator): Dietary intervention
  Interventions: Behavioral: SFA+Cys/Met diet

INTERVENTIONS:
Behavioral: PUFA-Cys/Met diet — Provision of food and supplements that are rich in polyunsaturated fatty acids (PUFA, n-3 and n-6) and low in the amino acids cysteine (Cys) and methionine (Met).
  Arms: Group A
Behavioral: SFA+Cys/Met diet — Provision of food and supplements that are rich in saturated fatty acids (SFA) and the amino acids cysteine (Cys) and methionine (Met).
  Arms: Group B

SUMMARY:
The aim of this study is to examine if changing stearoyl-coenzyme A desaturase-1 (SCD1) activity through dietary interventions can increase energy metabolism in humans.

DETAILED DESCRIPTION:
In rodents as well as humans, high stearoyl-coenzyme A desaturase-1 (SCD1) activity is considered to be involved in development of obesity. In animal models, polyunsaturated fatty acids (PUFA) inhibit Scd1 gene expression and at the population level, dietary PUFA and plasma PUFA show strong inverse associations with plasma SCD indices. Emerging evidence also suggests a role for the sulphur amino acid cysteine in regulating SCD1 activity and obesity.

The overall aim of the project is to examine if interventions that lowers SCD1 activity lead to increased energy metabolism. In this project, the investigators will conduct dietary intervention trials to evaluate the effects of short-term consumption of a diet rich in polyunsaturated fatty acids (PUFA) and low in cysteine and its precursor methionine (PUFA-Cys/Met) vs. a diet rich in saturated fatty acids (SFA) and cysteine/methionine (SFA+Cys/Met) on SCD1 activity, lipids, amino acids, glucose and other biomarkers related to energy metabolism, in healthy normal-weight subjects. Healthy volunteers will be randomized to the PUFA-Cys/Met or SFA+Cys/Met diets receiving supplements/meals in a single dose or for 7 days.

This study is a pilot study, with main focus on feasibility, tolerance and side effects. If the pilot shows positive results in terms of side effects, safety and tolerance, the investigators will follow-up by including obese subjects in a longer dietary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Healthy normal-weight (BMI 20-25 kg/m2)

Exclusion Criteria

* High physical activity
* Smoking
* High intake of fatty fish or cod liver oil
* Drugs
* Pregnancy or breastfeeding
* Chronic disease

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-02; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change in metabolic biomarkers | 0 hour and at 30 min, 1, 2, 3, 4, 6, 8, 12, 24, 48 and 72 h after single meal. Baseline and up to 7 days in 7 days intervention
  Measurement of biomarkers of amino acid and fatty acid metabolism, including plasma concentration of cysteine, methionine, fatty acids, and stearoyl CoA desaturase (SCD) indices

SECONDARY OUTCOMES:
Change in biomarkers of glucose metabolism | Baseline and up to 7 days
  Measurements of blood parameters including glucose and insulin, and Oral Glucose Tolerance Test
Change in biomarkers of triglycerides metabolism | Baseline and up to 7 days
  Measurements of blood parameters including LDL-/HDL-/VLDL-/total cholesterol, and triglycerides
Change in molecular signatures | Baseline and up to 7 days
  Evaluation of markers related to lipid, amino acid and glucose metabolism, including measurements of mRNA expression in blood cells, and proteins and metabolites, in blood and/or urine
Hunger and satiety patterns | Baseline and up to 7 days
  Evaluated by plasma levels of hormones such as leptin, ghrelin, cholecystokinin, GLP-1 and PYY
Appetite assessed by visual analogue scales | 0, 15, 30, 45, 60, 90, 120, 180 minutes postprandially (single meal intervention). Change from baseline up to 7 days (7 days intervention)
Change in inflammatory markers | Baseline and up to 7 days
  Measurements of blood parameters, e.g., CRP, cytokines and chemokines, adipokines, metabolic markers, hormones, growth factors, tissue remodeling proteins, angiogenesis markers, acute phase reactants, and other important circulating proteins.
Feasibility and compliance of the diet intervention | Up to 7 days
  Evaluated by compliance questionnaires
Tolerance of the diet intervention | Up to 7 days
  Assessed by blood pressure, pulse and laboratory parameters including haematology, clinical chemistry and urine analysis

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oslo, Oslo, Norway

REFERENCES:
- [Derived] Elshorbagy A, Bastani NE, Lee-Odegard S, Ovrebo B, Haj-Yasein N, Svendsen K, Turner C, Refsum H, Vinknes KJ, Olsen T. The association of fasting plasma thiol fractions with body fat compartments, biomarker profile, and adipose tissue gene expression. Amino Acids. 2023 Mar;55(3):313-323. doi: 10.1007/s00726-022-03229-2. Epub 2022 Dec 21. PMID 36542145
- [Derived] Olsen T, Ovrebo B, Turner C, Bastani NE, Refsum H, Vinknes KJ. Effects of short-term methionine and cysteine restriction and enrichment with polyunsaturated fatty acids on oral glucose tolerance, plasma amino acids, fatty acids, lactate and pyruvate: results from a pilot study. BMC Res Notes. 2021 Feb 2;14(1):43. doi: 10.1186/s13104-021-05463-5. PMID 33531059
- [Derived] Olsen T, Turner C, Ovrebo B, Bastani NE, Refsum H, Vinknes KJ. Postprandial effects of a meal low in sulfur amino acids and high in polyunsaturated fatty acids compared to a meal high in sulfur amino acids and saturated fatty acids on stearoyl CoA-desaturase indices and plasma sulfur amino acids: a pilot study. BMC Res Notes. 2020 Aug 10;13(1):379. doi: 10.1186/s13104-020-05222-y. PMID 32778150